CLINICAL TRIAL: NCT04980885
Title: A Phase Ib/II Trial of AK117 (Anti-CD47 Antibody) in Patients With Acute Myeloid Leukemia
Brief Title: A Trial of AK117 (Anti-CD47 Antibody) in Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK117-104
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK117+Azacitidine (Experimental): Phase Ib: Subjects will receive different doses of A117 in combination with azacitidine 75 mg/m2 subcutaneous daily for 7 days of a 28 day cycle;
  Phase II: Subjects will receive AK117 at the recommended Phase 2 dose in combination with azacitidine 75 mg/m2 subcutaneous daily for 7 days of a 28-day cycle.
  Interventions: Drug: AK117; Drug: Azacitidine

INTERVENTIONS:
Drug: AK117 — Subjects receive AK117 intravenously.
Drug: Azacitidine — Subjects receive Azacitidine subcutaneously.

SUMMARY:
This is a open label, phase Ib/II study. All patients are diagnosed with AML, Eastern Cooperative Oncology Group (ECOG) performance status 0-3. The purpose of this study is to evaluate the safety and efficacy of AK117 + azacitidine in subjects with AML.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3，and 0~2 are required for subjects ≥75 years old.
* Has a life expectancy of at least 12 weeks.
* Patient with AML diagnosed according to WHO 2016 criteria.
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Patient has acute promyelocytic leukemia.
* Patient has known active central nervous system (CNS) involvement with AML.
* Favorable risk cytogenetics such as t(8;21), inv(16) or t(16;16) or t(15;17) as per the National Comprehensive Cancer Network (NCCN) Guidelines Version 2, 2021 for AML.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has undergone major surgery within 30 days of Study Day 1.
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Previous allogeneic hematopoietic stem cell transplant (allo-HSCT) .
* Prior treatment with any anti-CD47 or anti-SIRPα (signal regulatory protein alpha) agent.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Patient with known allergy or hypersensitivity to AK117, azacitidine or any of their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission rate （complete remission + complete remission with incomplete count recovery） | Approximately 6 months
  Number of participants achieving a complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) per European LeukemiaNet (ELN) 2017 criteria.
Number of participants with adverse events (AEs) | Up to approximately 2 years.
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Rate of CR Without Minimal Residual Disease (CR MRD-) | Approximately 6 months
  The rate of CR MRD- is the percentage of participants who achieve a CR MRD- as defined by investigators based on ELN 2017 criteria.
Duration of complete response (DoCR) | Approximately 6 months
  The DoCR is measured from the time the assessment criteria are first met for CR (including CR MRD- and CR MRD+/unk) until the first date of AML relapse or death.
Overall Survival | Up to death or end of study
  The OS is measured from the date of treatment to the date of death from any cause.
Event-Free Survival (EFS) | Up to end of study
  The EFS is defined as time from the date of treatment to the earliest date of documented relapse from complete remission (CR), treatment failure , or death from any cause.
Maximum observed concentration (Cmax) of AK117 | Up to 2 years.
  Serum concentrations of AK117 in individual subjects at different time points after AK117 administration.
Anti-drug antibodies (ADA) | Up to 2 years.
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang, China